CLINICAL TRIAL: NCT06984835
Title: A Prospective, Multi-Center, Randomized, Controlled, Double-Blind, Split-Face Study of the Safety and Effectiveness of ELLANSÉ®-S Dermal Filler in the Treatment of Nasolabial Folds
Brief Title: Safety and Effectiveness of ELLANSÉ®-S Dermal Filler in the Treatment of Nasolabial Folds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AQTIS Medical B.V. (Other)
Collaborators: Sinclair Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SES001
Record Dates: First submitted 2025-04-28; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Nasolabial Folds
Keywords: nasolabial folds; NLF; NLFs; dermal filler; wrinkle; correction; wrinkles; Ellanse; Ellanse S; polycaprolactone; PCL; microspheres; resorbable

STUDY DESIGN:
Intervention Model Description: The study is a "split face" design; subjects will be treated in one nasolabial fold on one side of the face with one treatment device and with the comparator device in the nasolabial fold on the other side
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Ellanse S (Experimental): Polycaprolactone and carboxymethylcellulose gel based dermal filler
  Interventions: Device: Ellanse S
- Calcium Hydroxylapatite (Active Comparator): Calcium Hydroxylapatite and carboxymethylcellulose gel based dermal filler
  Interventions: Device: Calcium Hydroxylapatite-based filler

INTERVENTIONS:
Device: Ellanse S — Ellanse S polycaprolactone and carboxymethylcelluose gel based dermal filler syringe
  Arms: Ellanse S
Device: Calcium Hydroxylapatite-based filler — Calcium Hydroxylapatite and carboxymethylcellulose based filler
  Arms: Calcium Hydroxylapatite

SUMMARY:
The study will be a prospective, randomized, multi-center, split-face, controlled, double-blind clinical trial to evaluate the safety and effectiveness of ELLANSÉ®-S for the treatment of NLFs. Subjects will be randomized to receive treatment (ELLANSÉ®-S) in one NLF and control (Radiesse®) in the contralateral NLF. A total of 126 subjects will be treated. The control and test articles will be supplied in sterile ready-to-use, pre-filled syringes. Initial treatment and any 4-week touch-up will be done consistent with initial randomization. Any retreatment(s) in either NLF will be with ELLANSÉ®-S.

Subjects who meet Inclusion/Exclusion criteria will receive an initial treatment, an optional touch up at the 4-week visit, and may be eligible to receive retreatment at either 12 or 18 months after treatment (determined by when the fold has returned to baseline score, or the fold has lost at least 1 point on the Wrinkle Severity Rating Scale (WSRS) from optimal improvement). Retreatment to one side is allowed if only one side qualifies, but the other side may not be retreated at a later visit. If retreatment occurs, the subject may also be eligible to receive an optional touch up at the 4-week follow up visit. If a touch up occurs after the initial or retreatment injection, the subject will return for an additional safety visit 2 weeks after each injection. A week 4 safety visit will occur after retreatment touch-up. Primary effectiveness will be assessed at 6 months. All subjects will be followed for a minimum of 24 months after the initial treatment phase. After each injection, subjects will be contacted by telephone call/email after 72 hours and will return for a safety visit 2 weeks after treatment. At the week 4 visit, subjects will be assessed for a touch up. If a touch up is indicated as determined by the investigator, the investigator will use the same material as that used for initial treatment for the respective side. In addition, subjects will be seen at 6 weeks 3, 6, 9, 12, 18, and 24 months (from the end of the initial treatment phase). Subjects receiving a retreatment (at 12 or 18 months after treatment) will return for additional safety visits at 2 weeks and 3 and 6 months after this retreatment (the 6 month coincides with regularly scheduled visit). Subjects will have the option of a retreatment touch up injection at 4 weeks after retreatment, and if they do will have another call at 72hrs and a week 2 safety visit.

The validated Wrinkle Severity Rating Scale will be used for assessment of the primary effectiveness endpoint (1). Assessment of the secondary effectiveness endpoints will include use of WSRS, the Global Aesthetic Improvement Scale (GAIS), VAS pain assessment, the validated FACE-Q Appraisal of Nasolabial Folds Questionnaire, the FACE-Q Satisfaction with Treatment Outcome Scale and the FACE-Q Age Appraisal VAS.

The study will last approximately 30 months. All subjects will be recruited within approximately 6 months after the recruitment of the first subject and followed for a minimum of 24 months after the initial treatment visit. Subjects receiving a retreatment (at 12 or 18 months) will receive a telephone call/email 72 hours after retreatment and they will return for an additional safety visit 2 weeks after retreatment. Subjects may receive a retreatment touch up at 4 weeks after retreatment, and if touched up, will have safety visits at 2 and 4 weeks. All retreated subjects will also be asked to attend month 3 and month 6 safety visits. The 6-month safety visit will correspond with the next study visit (e.g., 18 month or 24-month visit depending on when they are reinjected)

126 male and female subjects will be enrolled. This enrollment number accounts for a 20% attrition rate, to ensure an adequate safety population for long-term follow-up, and a Per Protocol Set (PPS) of at least 101 NLFs per treatment arm. At least 20% of treated subjects will have Fitzpatrick Skin Types IV, V, and VI. Of these, at least, 10% will be Type IV, 5% Type V and 5% Type VI. The investigative sites will be encouraged to enroll both male and female subjects. In addition, up to 2 non-randomized, non-split-face run-in subjects will be treated with ELLANSÉ®-S by each investigator to allow the investigator to become familiar with injection characteristics. This run-in cohort will be required to meet all study inclusion/exclusion criteria and will be followed in the same manner as the non-run-in cohort. Up to seven US sites will participate.

ELIGIBILITY:
Inclusion Criteria:

Only subjects meeting all of the following inclusion criteria will be considered for study enrollment:

1. Subject is male or female aged at least 22 years.
2. Subject has bilateral moderate or severe (symmetric grade 3 or 4) NLFs on the WSRS as scored by the treating investigator.
3. Subject is willing to abstain from other facial aesthetic procedures in the lower face including the NLFs through the study period (up to the final follow-up visit, depending on retreatment) which could interfere with treatment outcomes (e.g. facial fillers, skin laser and radiofrequency therapy such as Thermage, chemical re-surfacing, dermabrasion, Botox injections, aesthetic facial surgery, other facial treatments in the NLFs).
4. Subject understands and accepts the obligation to present for all scheduled follow-up visits and is logistically able to meet all study requirements.
5. Subject with facial hair which may obstruct the assessment of the treatment area, must be agreeable with non-laser removal of facial hair prior to assessment visits.
6. Subject agrees to avoid dental procedures (surgery, implants, dental work) for 3 weeks after any treatment.
7. Subject is willing to provide written informed consent for their participation in the study.
8. Subject has best corrected visual acuity of 20/40 or better (in each eye), and have normal confrontational visual fields, and normal extraocular motility.

Exclusion Criteria:

Subjects having any of the following criteria, either at screening or at baseline, will not be included in the study:

1. Subject is a female of childbearing potential (e.g., not postmenopausal for at least one year or has not had a hysterectomy or tubal ligation) not using medically effective birth control (e.g., hormonal methods in use at least 30 days prior to injection or barrier methods such as condom and spermicide in use at least 14 days prior to injection) or is pregnant, lactating, or plans to become pregnant during the study.
2. Subject has participated in a clinical study in which an investigational device or drug was received in the 30 days prior to screening or plans to enroll in such a study during the course of the current study.
3. Subject is an employee or direct relative of an employee of the investigational site or study sponsor.
4. Subject has received surgery in the NLFs.
5. Subject has received facial threads or autologous fat injections in the face.
6. Subject has a serious or progressive disease, which, in the investigator's judgment, puts the subject at undue risk (e.g., uncontrolled diabetes, autoimmune disease, cardiac pathologies).
7. Subject has an acute inflammatory process or infection, or history of chronic or recurrent infection or inflammation with the potential to interfere with the study results or increase the risk of adverse events.
8. Subject has a disorder that may impact wound healing such as connective tissue or immunosuppressive disorder.
9. Subject has a history of precancerous lesions/skin malignancies.
10. Subject has had an active skin disease within the past 6 months.
11. Subject has scars, infection, rosacea, herpes, acne, blotches or other pathology in the NLFs that in the Investigator's opinion will affect evaluation or treatment.
12. Subject has facial hair covering the nasolabial folds that they are unwilling to remove for study assessments.
13. Subject has a past history of systemic streptococcal disease or an active streptococcus infection.
14. Subject has had a COVID-19 vaccine within 2 weeks of scheduled injections or plans to receive one 3 weeks after any study injection.
15. Subject was ill with a virus (SARS, COVID, flu) within 2 weeks of scheduled injection.
16. Subject is predisposed to keloidosis or hypertrophic scarring.
17. Subject has a known history of hyper- or hypo-pigmentation in the NLFs.
18. Subject with known allergy to poly (ε-caprolactone), phosphate buffered saline, glycerine, calcium hydroxylapatite (CaHA), or sodium carboxymethylcellulose.
19. Subject has a known history of multiple allergies, allergic/anaphylactic reactions including hypersensitivity to lidocaine or anesthetics of the amide type.
20. Subject has a known bleeding disorder.
21. Subject has received within the past 2 weeks or plans to receive up to 1 week after treatment high-dose Vitamin E, aspirin, anti-inflammatories, antiplatelets, thrombolytics or any other medication that could increase the risk of bleeding.
22. Subject has received any medication which, in the judgement of the investigator, may interfere with the study objectives.
23. Subject has received within the past 12 months or plans to receive during the study any injections outside of those in the study protocol including non-permanent fillers (e.g., hyaluronic acid) or neurotoxin on the face below cheekbone (forehead is acceptable).
24. Subject has received at any time or plans to receive during the study a permanent filler (e.g., PMMA, silicone) on the face below the cheekbone.
25. Subject has received within the past 24 months or plans to receive during the study a semi-permanent or long last filler (e.g. polylactic acid or calcium hydroxylapatite CaHA) on the face.
26. Subject has received within the past 6 months or plans to receive during the study dermal resurfacing procedures or non-invasive skin tightening or energy based or mechanical or chemical aesthetic procedure on the face.
27. Subject has received in the past 4 weeks or plans to receive during the study prescription facial wrinkle therapies (tretinoin), topical steroids,
28. Subject has received within the past 2 weeks skin irritating topical preparations, or self-tanning agents on the face.
29. Subject has received within the past 6 months systemic retinoids.
30. Subject has received within the past 3 months systemic steroids or chemotherapy or immunosuppressive agents.
31. Subject has a known history of ongoing rapid weight loss/gain or plans to begin a weight loss program during the study (5% of body weight).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean Change in NLF WSRS score from baseline at 6 months by a live, masked reviewer | 6 months
  The primary effectiveness endpoint uses the 6-month and baseline Wrinkle Severity Rating Scale (WSRS) scores as determined by a live, masked reviewer. The change from baseline on the WSRS at 6 months of NLFs in the ELLANSÉ®-S treatment arm will be compared to that of NLFs in the Radiesse® control arm. The statistical objective is to demonstrate non-inferiority of WSRS improvement in the NLF indication of ELLANSÉ®-S to Radiesse®.
  Note: the WSRS provides 5 scoring options from 1 Absent to 5 Extreme. A lower score is a better clinical outcome.

SECONDARY OUTCOMES:
Difference in mean change from baseline on the Wrinkle Severity Rating Scale (WSRS) at 12 months as rated by a live, masked reviewer | 12 months
  Difference in mean change from baseline on the Wrinkle Severity Rating Scale (WSRS) at 12 months as rated by a live, masked reviewer Note: the WSRS provides 5 scoring options from 1 Absent to 5 Extreme. A lower score is a better clinical outcome.
Global Aesthetic Improvement Scale (GAIS) response rate at 6 months as rated by the live, masked reviewer | 6 months
  Global Aesthetic Improvement Scale (GAIS) response rate at 6 months as rated by the live, masked reviewer Note: There are 5 scoring options ranging from from "Very Much Improved" to "Worse"
Difference in mean change in total score on the FACE-Q Appraisal of Nasolabial Folds Questionnaire at 6 months. | 6 months
  Difference in mean change in total score on the FACE-Q Appraisal of Nasolabial Folds Questionnaire at 6 months.
  Note: 4 responses can be chosen; not at all (1), a little (2), moderately (3) and extremely (4), a lower score is a better clinical outcome
Difference in mean change in total score on the FACE-Q Appraisal of Nasolabial Folds Questionnaire at 12 months | 12 months
  Difference in mean change in total score on the FACE-Q Appraisal of Nasolabial Folds Questionnaire at 12 months.
  Note: 4 responses can be chosen; not at all (1), a little (2), moderately (3) and extremely (4), a lower score is a better clinical outcome
Difference in mean change from baseline on the Wrinkle Severity Rating Scale (WSRS) at 18 months as rated by a live, masked reviewer. | 18 months
  Difference in mean change from baseline on the Wrinkle Severity Rating Scale (WSRS) at 18 months as rated by a live, masked reviewer.
  Note: the WSRS provides 5 scoring options from 1 Absent to 5 Extreme. A lower score is a better clinical outcome.
Individual endpoints at each time point of, 6 weeks, 3, 6, 9, 12, and 18, and 24 months for responders on the Wrinkle Severity Rating Scale (WSRS), as determined by a live, masked reviewer.ry Endpoint 1 | 6 weeks, 3, 6, 9, 12, 18 and 24 months
  Individual endpoints at each time point of, 6 weeks, 3, 6, 9, 12, and 18, and 24 months for responders on the Wrinkle Severity Rating Scale (WSRS), as determined by a live, masked reviewer.
  Note: the WSRS provides 5 scoring options from 1 Absent to 5 Extreme. A lower score is a better clinical outcome.
Individual endpoints at each time point of 6 weeks, 3, 9, and 24 months for change from baseline on the Wrinkle Severity Rating Scale (WSRS), as determined by a live, masked reviewer. | 6 weeks, 3, 9 and 24 months
  Individual endpoints at each time point of 6 weeks, 3, 9, and 24 months for change from baseline on the Wrinkle Severity Rating Scale (WSRS), as determined by a live, masked reviewer.
  Note: the WSRS provides 5 scoring options from 1 Absent to 5 Extreme. A lower score is a better clinical outcome.
Individual endpoints at 6 weeks, 3, 6, 9, 12, 18, & 24 months for the comparative improvement on the Wrinkle Severity Rating Scale (WSRS) by subject of NLFs in the ELLANSÉ®-S arm to NLFs in the Radiesse® arm, as determined by a live, masked evaluator | 6 weeks, 3, 6, 9, 12, 18 and 24 months
  Individual endpoints at each time point of 6 weeks, 3, 6, 9, 12, 18, and 24 months for the comparative improvement on the Wrinkle Severity Rating Scale (WSRS) by subject of NLFs in the ELLANSÉ®-S treatment arm to NLFs in the Radiesse® arm, as determined by a live, masked evaluator.
  Note: the WSRS provides 5 scoring options from 1 Absent to 5 Extreme. A lower score is a better clinical outcome.
Individual endpoints at each time point of 6 weeks, 3, 6, 9, 12, 18, and 24 months for change from baseline on the Wrinkle Severity Rating Scale (WSRS), as determined by a blinded photographic review panel | 6 weeks, 3, 6, 9, 12, 18 and 24 months
  Individual endpoints at each time point of 6 weeks, 3, 6, 9, 12, 18, and 24 months for change from baseline on the Wrinkle Severity Rating Scale (WSRS), as determined by a blinded photographic review panel.
  Note: the WSRS provides 5 scoring options from 1 Absent to 5 Extreme. A lower score is a better clinical outcome.
Individual endpoints at 6 weeks, 3, 6, 9, 12, 18, & 24 months for the proportion of NLFs in the ELLANSÉ®-S arm compared to NLFs in the Radiesse® arm with ≥1 point improvement from baseline on the WSRS as determined by a blinded photographic review panel | 6 weeks, 3, 9, 12, 18 and 24 months
  Individual endpoints at each time point of 6 weeks, 3, 6, 9, 12, 18, and 24 months for the proportion of NLFs in the ELLANSÉ®-S treatment arm compared to that of NLFs in the Radiesse® arm with ≥1 point improvement from baseline on the Wrinkle Severity Rating Scale (WSRS), as determined by a blinded photographic review panel.
  Note: the WSRS provides 5 scoring options from 1 Absent to 5 Extreme. A lower score is a better clinical outcome.
Individual endpoints at each time point of 6 weeks, 3, 6, 9, 12, 18, and 24 months for GAIS scores for ELLANSÉ®-S and Radiesse®. Individual endpoints for each rater type, as rated by: 1) Live masked evaluator 2) Treating investigator 3) The study subject | 6 weeks, 3, 6, 9, 12, 18 and 24 months
  Individual endpoints at each time point of 6 weeks, 3, 6, 9, 12, 18, and 24 months for GAIS scores for ELLANSÉ®-S and Radiesse®. Individual endpoints for each rater type, as rated by:
  * Live, masked evaluator (excluding the 6 month),
  * treating investigator;
  * and the study subject.
Individual endpoints at each time point of 6 weeks, 3, 9, 18, and 24 months for change from baseline for ELLANSÉ®-S and Radiesse® on the Subject FACE-Q Appraisal of Nasolabial Folds Questionnaire | 6 weeks, 3, 9, 12, 18 and 24 months
  Individual endpoints at each time point of 6 weeks, 3, 9, 18, and 24 months for change from baseline for ELLANSÉ®-S and Radiesse® on the Subject FACE-Q Appraisal of Nasolabial Folds Questionnaire.
  Note: 4 responses can be chosen; not at all (1), a little (2), moderately (3) and extremely (4), a lower score is a better clinical outcome
Individual endpoints at each time point of 6 and 12 months for change from baseline for ELLANSÉ®-S and Radiesse® on the Subject FACE-Q Satisfaction with Outcome Scale | 6 and 12 months
  Individual endpoints at each time point of 6 and 12 months for change from baseline for ELLANSÉ®-S and Radiesse® on the Subject FACE-Q Satisfaction with Outcome Scale.
  Note: 4 responses can be chosen; definitely disagree (1), somewhat disagree (2) somewhat agree (3) and definitely agree (4); a higher score is a better clinical outcome
Visual Analogue Scale (VAS) pain assessment in NLFs treated with ELLANSÉ®-S compared to NLFs treated with Radiesse® at initial injection | Baseline, 4 week post injection touch up visits, optional 12 month retreatment, optional 18 month retreatment
  Visual Analogue Scale (VAS) pain assessment in NLFs treated with ELLANSÉ®-S compared to NLFs treated with Radiesse® at initial injection.
  Note: the scale ranges from 0 - no pain to 10 - worst pain with 0.5 point increments
Duration of treatment effect as measured on the Wrinkle Severity Rating Scale (WSRS) by ≥1 point improvement, for those NLFs that did not receive retreatment prior to the assessment time point at 18 and 24 months. | 18 and 24 months
  Duration of treatment effect as measured on the Wrinkle Severity Rating Scale (WSRS) by ≥1 point improvement, for those NLFs that did not receive retreatment prior to the assessment time point at 18 and 24 months.
  Note: the WSRS provides 5 scoring options from 1 Absent to 5 Extreme. A lower score is a better clinical outcome.
  Time Frame: 6 weeks, 3, 9, 12, 18 and 24 months
Duration of treatment effect as measured on the Wrinkle Severity Rating Scale (WSRS) by ≥1 point improvement, for those NLFs that did not receive retreatment prior to the assessment time point at 18 and 24 months. | Up to 24 months
  Time until return to baseline on the Wrinkle Severity Rating Scale (WSRS) for NLFs in the ELLANSÉ®-S treatment arm compared to that of NLFs in the Radiesse® arm.
  Note: the WSRS provides 5 scoring options from 1 Absent to 5 Extreme. A lower score is a better clinical outcome.

OTHER OUTCOMES:
The safety endpoint is to assess the rate and severity of adverse events from initial treatment through last study visit | Through to 24 months
  The safety endpoint is to assess the rate and severity of adverse events from initial treatment through last study visit. All AEs that occur throughout the duration of the study will be captured. Adverse events will be categorized by type, duration, severity, relationship to the study device and need for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy B Green, Principal Investigator — Skin Research Institute LLC
Locations (7):
- United States (7):
  - Investigate MD, Scottsdale, Arizona
  - Clinical Testing of Beverly Hills, Encino, California
  - DMR Research, PLLC, Westport, Connecticut
  - Skin Research Institute LLC, Miami, Florida
  - Callender Center for Clinical Research, Glenn Dale, Maryland
  - Skincare Physicians, Chestnut Hill, Massachusetts
  - Advanced Dermatology of Michigan, Warren, Michigan

IPD SHARING:
Plan to Share IPD: Undecided